CLINICAL TRIAL: NCT00547443
Title: A Randomized Phase I/II Study Of Sorafenib In Combination With High Does Chemoradiation In Patients With Stage IIIA/B Non-small Cell Lung Cancer (NSCLC)
Brief Title: Sorafenib and High-Dose Carboplatin, Paclitaxel, and External-Beam Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn as the sponsor has stopped the drug for NSCLC population
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-03507; SCCC-052007-068; BAYER-SCCC-052007-068; CDR0000571535 (Registry Identifier: PDQ (Physician Data Query)); NCT00975260 (obsolete NCT alias)
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer; large cell lung cancer; bronchoalveolar cell lung cancer; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Paclitaxel; Sorafenib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Active Comparator): Patients receive chemoradiotherapy comprising paclitaxel, carboplatin, and high-dose external beam radiotherapy (HDRT) as in phase I. Patients also receive consolidation therapy comprising paclitaxel and carboplatin as in phase I.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy
- Arm II (Experimental): Patients receive chemoradiotherapy comprising paclitaxel, carboplatin, and HDRT as in phase I. Patients also receive consolidation therapy comprising paclitaxel, carboplatin, and sorafenib tosylate at the MTD as in phase I, as well as maintenance therapy comprising sorafenib tosylate at the MTD as in phase I.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: sorafenib tosylate; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: paclitaxel — Given IV
Drug: sorafenib tosylate — Given orally
  Arms: Arm II
Radiation: radiation therapy — Given 5 days a week for 7.5 weeks

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving sorafenib together with high-dose chemotherapy and external-beam radiation therapy may kill more tumor cells.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of sorafenib when given together with high-dose carboplatin, paclitaxel, and external-beam radiation therapy in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the median survival from randomization for patients receiving carboplatin and paclitaxel with high-dose radiation therapy (HDRT) or same regimen with sorafenib tosylate.

Secondary

* To determine the overall response rate, failure-free survival, and survival for patients receiving carboplatin/paclitaxel with 74 Gy HDRT or same regimen with sorafenib tosylate.
* To determine the feasibility of concurrent sorafenib tosylate and chemoradiation as measured by safety (the rate of grade 3 or higher radiation related esophagitis or pulmonary toxicity or chemotherapy related grade 4 hematological or other non-hematological toxicities occurring within 60 days of the start of treatment) and compliance (the completion of the treatment regimen with no more than minor variations).
* To correlate outcomes (survival, toxicity, quality of life) with biological parameters.

OUTLINE: This is a multicenter study.

* Phase I:

  * Chemoradiotherapy: Patients receive paclitaxel IV over 60 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats weekly for 7 weeks. Patients undergo concurrent high-dose external beam radiotherapy (HDRT) 5 days a week for 7.5 weeks. Cohorts of patients also receive escalating doses of oral sorafenib tosylate twice daily for 7 weeks.
  * Consolidation therapy: Beginning at week 11, patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 6 weeks. Patients also receive oral sorafenib tosylate at the maximum tolerated dose (MTD) twice daily.
  * Maintenance: Patients receive oral sorafenib tosylate twice daily at the MTD.
* Phase II: Patients are randomized to 1 of 2 treatment arms.

  * Arm I:

    * Chemoradiotherapy: Patients receive paclitaxel, carboplatin, and HDRT as in phase I.
    * Consolidation therapy: Patients receive paclitaxel and carboplatin as in phase I.
  * Arm II:

    * Chemoradiotherapy: Patients receive paclitaxel, carboplatin, and HDRT as in phase I. Patients also receive oral sorafenib tosylate as in phase I at the MTD.
    * Consolidation therapy: Patients receive paclitaxel, carboplatin, and sorafenib tosylate at the MTD as in phase I.
    * Maintenance: Patients receive sorafenib tosylate at the MTD as in phase I. After completion of study therapy, patients are followed every 3 months for 2 years and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically documented non-small cell lung cancer (NSCLC)

  * Any of the following subtypes allowed:

    * Adenocarcinoma (including bronchoalveolar cell)
    * Squamous cell carcinoma
    * Large cell anaplastic carcinoma (including giant and clear cell carcinomas)
    * Poorly differentiated (not otherwise specified) NSCLC
  * No metastasis (patients must be M0)
  * Stage IIIA (T1 or T2 with N2 or T3N1-2) or stage IIIB (T4 with any N or any T with N2 or N3) disease
* Measurable disease
* Tumors adjacent to a vertebral body are allowed as long as all gross disease can be encompassed in the radiation boost field

  * The boost volume must be limited to < 50% of the ipsilateral lung volume
* Pleural effusion that is a transudate, cytologically negative, and nonbloody allowed if the radiation oncologists feel the tumor can still be encompassed within a reasonable field of radiotherapy

  * Pleural effusions seen on the chest CT but too small to tap allowed

Exclusion criteria:

* Totally resected tumors
* Exudative, bloody, or cytologically malignant effusions
* Known brain metastasis

  * Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Zubrod performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL (prior to transfusions)
* Total bilirubin ≤ 1.5 mg/dL
* AST or ALT ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Glucose ≤ 2 times ULN
* Creatinine ≤ 2.0 mg/dL
* FEV_1 ≥ 1,200 mL
* Weight loss ≤ 10% over the past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Women of childbearing potential and male participants who are unwilling or unable to use an acceptable method of contraception throughout the study and for 4 weeks after completion of treatment or those who are using a prohibited contraceptive method
* INR < 1.5 or a PT/PTT within normal limits

Exclusion criteria:

* Known allergy to murine proteins or Cremophor EL
* Active pulmonary infection not responsive to conventional antibiotics
* History of severe chronic obstructive pulmonary disease requiring ≥ 3 hospitalizations over the past year
* Cardiac disease including any of the following:

  * Congestive heart failure > class II NYHA
  * Unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months)
  * Myocardial infarction within the past 6 months
  * Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Patients with neuropathy > grade 1
* Evidence of malignancy in the past 2 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other in situ cancer
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management
* Known HIV infection or chronic hepatitis B
* Active clinically serious infection > CTCAE grade 2
* Thrombolic or embolic events, such as a cerebrovascular accident including transient ischemic attacks, within the past 6 months
* Pulmonary hemorrhage or bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* Any other hemorrhage or bleeding event ≥ CTCAE Grade 3 within the past 4 weeks
* Serious nonhealing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Known or suspected allergy to sorafenib tosylate or any agent given in the course of this trial
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem
* Significant traumatic injury within the past 4 weeks

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Recovered from exploratory thoracotomy
* Concurrent anti-coagulation treatment with an agent such as warfarin or heparin allowed provided INR or PT/PTT requirements are met

Exclusion criteria:

* Prior systemic chemotherapy for lung cancer and/or thoracic/neck radiotherapy for any reason
* Prior surgical resection of present cancer
* Prior therapy with any molecular-targeted drugs (for lung cancer)
* Currently participating in other phase III therapeutic clinical trials and/or who have participated in other phase III therapeutic clinical trials in the previous 30 days
* Major surgery or open biopsy within the past 4 weeks
* Concurrent Hypericum perforatum (St. John's wort) or rifampin (rifampicin)
* Other concurrent anticancer drugs, including hormonal, immunotherapeutic, or chemotherapeutic agents

  * Steroids for acute symptom management, adrenal failure, septic shock, or as antiemetics allowed
  * Hormones administered for nondisease-related conditions (e.g., insulin for diabetes) allowed
* Amifostine concurrently with radiotherapy or within 3 months of completion of radiotherapy
* Concurrent colony-stimulating factors (i.e., filgrastim [G-CSF] or sargramostim [GM-CSF])

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Median survival | Mean 24-Months
  To determine the median survival from randomization for patients receiving carboplatin / paclitaxel with high dose radiation therapy or same regimen with Sorafenib.

SECONDARY OUTCOMES:
Progression-free survival | Mean 24-Months
  To determine the overall response rate, failure-free survival and survival for patients receiving carboplatin / paclitaxel with high dose radiation therapy or same regimen with Sorafenib.

CONTACTS AND LOCATIONS:
Overall Officials: Hak Choy, MD, Study Chair — Simmons Cancer Center
Locations (2):
- United States (2):
  - Arlington Cancer Center - Arlington, Arlington, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas